CLINICAL TRIAL: NCT01757886
Title: inflAmmatory maRkers in Blood and Thrombus Aspirated From Patients With acutE myocaRdial Infarction With St-segment elevAtion
Acronym: ARTERIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Responsible Party: Principal Investigator, Enrique Quintero, Alberto Dominguez Rodriguez, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Other Study IDs: ARTERIA-2012; ARTERIA-2012 (Other: Fundacion Canaria Rafael Clavijo)
Record Dates: First submitted 2012-12-22; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Patients Admitted With the Diagnosis of ST-elevation Acute Coronary Syndrome
Keywords: Myocardial infarction, Inflammation, Thrombus, Coronary angioplasty.
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

GROUPS / COHORTS (1):
- ST-elevation acute coronary syndrome: ARTERY is a prospective, multicenter, which will include patients admitted with the diagnosis of ST-elevation acute coronary syndrome and thrombus aspiration is performed during primary angioplasty
  Interventions: Other: Biomarkers to analyze both intracoronary thrombi as blood

INTERVENTIONS:
Other: Biomarkers to analyze both intracoronary thrombi as blood

SUMMARY:
The prognostic value of inflammatory markers in acute coronary syndrome has been extensively demonstrated, however it is still unknown whether there is an association between circulating and local (thrombus) inflammatory molecules, and the subset of molecules that provide better prognostic information in patients with ST-elevation acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* They include patients of both sexes, without limits of age, with a diagnosis of STEMI within 12 hours after the beginning of symptoms. ST-elevation myocardial infarction was defined in the presence of symptoms consistent, persistent elevation (> 20 min) ST segment ≥ 1 mm in at least two contiguous leads or in the presence of left bundle branch block presumably new onset and cardiac troponin I elevation

Exclusion Criteria:

* Injury significant common core of left coronary artery (stenosis greater than or equal to 50% of the vessel lumen).
* Pre-Fibrinolysis percutaneous coronary intervention.
* Previous coronary bypass surgery.
* Thyrotoxicosis.
* Having an inflammatory systemic or local inflammatory process.
* Malignant neoplasm.
* Any disease that seriously compromise the prognosis and / or systemic inflammatory response generated.
* No thrombotic material obtained in the thrombus or insufficient for performing biochemical determinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pilot, prospective cohort, which included all patients admitted with a diagnosis of ST-elevation myocardial infarction and undergoing thrombus aspiration during a procedure effective emerging percutaneous coronary revascularization.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to find out whether there is an association between certain inflammatory markers in blood and intracoronary thrombus and whether these markers are associated with the composite of all-cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Dominguez-Rodriguez, MD, PhD, Study Chair — Hospital Universitario de Canarias
Locations (2):
- Spain (2):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife